CLINICAL TRIAL: NCT06136689
Title: Role of Aortic Valve Composition in Pathophysiology and Diagnosis of Aortic Stenosis
Acronym: COMP-AS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University of Warsaw (Other)
Collaborators: Polish Cardiac Society (Other)
Responsible Party: Principal Investigator, Kajetan Grodecki, Principal Investigator, Medical University of Warsaw
Other Study IDs: 1WR/DAR15
Record Dates: First submitted 2023-11-07; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Aortic Stenosis; Aortic Valve Disease; Aortic Valve Calcification
MeSH Terms: conditions — Aortic Valve Stenosis; Aortic Valve Disease; Aortic Valve, Calcification of

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — leaflets of each aortic valve excised at the time of surgery will be separately placed in a pre-filled container with 10% neutral, phosphate-buffered formalin
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Severe Aortic Stenosis - High Flow, High Gradient: patients undergoing surgical aortic valve replacement for severe AS
- Severe Aortic Stenosis - classical Low Flow, Low Gradient: patients undergoing surgical aortic valve replacement for severe AS
- Severe Aortic Stenosis - paradoxical Low Flow, Low Gradient: patients undergoing surgical aortic valve replacement for severe AS
- Moderate Aortic Stenosis: patients undergoing aortic root replacement (Bentall procedure)
- Heart Transplant: patients undergoing orthotopic heart transplant for any reason

SUMMARY:
The study aims to evaluate composition differences of aortic valves in different stages and phenotypes of aortic stenosis using non-invasive imaging and histology.

ELIGIBILITY:
Inclusion Criteria:

* aortic valve replacement or heart transplant as part of standard care decided by the local Heart Team
* pre-surgical computed tomography angiography
* informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will involve patients undergoing surgical aortic valve replacement (SAVR) for different phenotypes of severe AS (high-flow high-gradient, classical low-flow low-gradient, and paradoxical low-flow low-gradient) or moderate AS with coexisting aortic aneurysm as part of Bentall procedure. Patients undergoing heart transplant will be considered control group without aortic valve stenosis.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Aortic valve tissue composition measured from pre-procedural computed tomography angiography | up to 30-days before surgery
  Quantitative analysis of aortic valve composition will be based on pre-surgical planning CTA images using semi-automated software (Autoplaque version 2.5, Cedars-Sinai Medical Center, Los Angeles, CA, USA) for calcified, non-calcified and total tissue volumes.
Aortic valve tissue composition measured from quantitative histology | immediately post-surgery
  Different stains will be used to characterize composition of excised aortic valves (hematoxylin and eosin, Movat Pentachrome, Van Gieson's trichrome, Congo Red, anti-CD68 antibody

CONTACTS AND LOCATIONS:
Overall Officials: Zenon Huczek, MD,PhD, Study Director — Medical University of Warsaw
Locations (2):
- Poland (2):
  - Medical University of Silesia, Katowice
  - Poznan University of Medical Sciences, Poznan

REFERENCES:
- [Background] Grodecki K, Tamarappoo BK, Huczek Z, Jedrzejczyk S, Cadet S, Kwiecinski J, Rymuza B, Parma R, Olasinska-Wisniewska A, Fijalkowska J, Protasiewicz M, Walczak A, Nowak A, Gocol R, Slomka PJ, Reczuch K, Jagielak D, Grygier M, Wojakowski W, Filipiak KJ, Dey D. Non-calcific aortic tissue quantified from computed tomography angiography improves diagnosis and prognostication of patients referred for transcatheter aortic valve implantation. Eur Heart J Cardiovasc Imaging. 2021 May 10;22(6):626-635. doi: 10.1093/ehjci/jeaa304. PMID 33247903